CLINICAL TRIAL: NCT06015178
Title: A Superiority Randomized Controlled Trial of the Effect of a Novel Intelligent Language Model on the Self-learning Ability of Medical Researchers
Brief Title: Enhancing Medical Researchers' Self-learning With an Intelligent Language Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023KYPJ222
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Medical Artificial Intelligence; Interdisciplinary Research; Self-Directed Learning
Keywords: medical artificial intelligence; Large Language Model; superiority randomized controlled trial; Self-Directed Learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent Language Model Group (Experimental): Subjects must use the intelligent language model to complete the retrieval and protocol design execution of an interdisciplinary task, in addition to Google search, literature search and book query.
  Interventions: Other: Intelligent Language Model
- Control Group (Placebo Comparator): Subjects can only use Google search, literature retrieval and book query, and cannot use any AI-driven conversational natural language processing tools to complete the retrieval and protocol design execution of an interdisciplinary task.
  Interventions: Other: control

INTERVENTIONS:
Other: Intelligent Language Model — Subjects must use the intelligent language model to complete the retrieval and protocol design execution of an interdisciplinary task, in addition to Google search, literature search and book query.
  Arms: Intelligent Language Model Group
Other: control — Subjects can only use Google search, literature retrieval and book query, and cannot use any AI-driven conversational natural language processing tools to complete the retrieval and protocol design execution of an interdisciplinary task.
  Arms: Control Group

SUMMARY:
Solving medical scientific problems is a crucial driving force behind the advancement of medical disciplines. As the complexity of scientific questions increases, an increasing number of problems require interdisciplinary collaboration to be resolved. However, most medical researchers lack interdisciplinary background knowledge and require substantial time to systematically learn relevant knowledge and skills. Furthermore, the continuous emergence of new knowledge and skills emphasizes the importance of researchers' ability for autonomous learning in the medical field. Therefore, to promote the development of medical disciplines, there is an urgent need for an effective method to enhance researchers' self-directed learning abilities for conducting interdisciplinary research.

The next-generation artificial intelligence language models, exemplified by ChatGPT, hold great potential in assisting researchers to access knowledge and information from various domains. Whether researchers can leverage such AI tools to enhance their self-directed learning abilities for conducting interdisciplinary research remains to be further explored. Additionally, concerns have been raised regarding the potential degradation of cognitive abilities through their use, although valid evidence is currently lacking.

To investigate whether AI tools, represented by ChatGPT, can effectively assist medical researchers in conducting interdisciplinary research and whether their usage may negatively impact researchers' cognitive abilities, a randomized controlled trial is warranted. This trial aims to ascertain the potential benefits and risks associated with utilizing AI tools in the medical research domain.

ELIGIBILITY:
Inclusion Criteria:

* Junior ophthalmologist with 1-3 years of clinical experience
* 20-28 years old, regardless of gender
* No prior experience in interdisciplinary research involving digital medicine
* Self-reported a minimum of 20 hours of participation in this study during the trial period
* Agree to participate in this study and sign informed consent

Exclusion Criteria:

* Individuals with reading difficulties or reading disabilities
* Reluctance to participate in this study

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
completion rate | through study completion, an average of 9 months
  The number of people who completed the task within the given time / the total number of people in the group

SECONDARY OUTCOMES:
Feasibility of the research program | through study completion, an average of 9 months
  The feasibility of the scheme is scored by a scoring group composed of experts. The feasibility is divided into 1-5 points according to the correctness and integrity of the key steps and details of the test. The higher the score, the higher the feasibility. The 1 point represents more than half of the key steps are missing or wrong, and the 5 point represents all the key steps and the details are appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shang Y, Lin Y, Li R, Shang Y, Li M, Zhao L, Jin L, Xu A, Liu D, Wu Q, Luo M, Pang J, Bi S, He Y, Xu M, Chen X, Cao Z, Yu S, Zhao J, Lai Y, Chen W, Lin H. The effectiveness of large language models in medical AI research for physicians: A randomized controlled trial. Cell Rep Med. 2025 Dec 16;6(12):102469. doi: 10.1016/j.xcrm.2025.102469. Epub 2025 Nov 26. PMID 41308643